CLINICAL TRIAL: NCT01609166
Title: Placebo-controlled Trial to Determine the Effectiveness of a 3% Allopurinol-base Topical Agent for Prevention of Capecitabine-induced Hand-foot Syndrome
Brief Title: Effectiveness Allopurinol Topical Agent Prevention Capecitabine-induced Hand-foot Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: IIB-ALO-2010-02; 2010-022095-31 (EudraCT Number)
Record Dates: First submitted 2012-05-24; First posted 2012-05-31 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2014-05

CONDITIONS: Hand-foot Syndrome
Keywords: Hand-foot Syndrome; capecitabine; allopurinol
MeSH Terms: conditions — Hand-Foot Syndrome | interventions — Allopurinol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Allopurinol 3% cream (Experimental): Allopurinol 3% cream in one side of the body
  Interventions: Drug: Allopurinol
- Placebo cream (Placebo Comparator): Placebo cream in the other side of the body
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Allopurinol — Allopurinol 3% cream application in one side of the body, twice a day for 6 months
  Arms: Allopurinol 3% cream
Drug: Placebo — Placebo cream application in the other side of the body, twice a day for 6 months
  Arms: Placebo cream

SUMMARY:
Hand-foot syndrome (HFS) is a dose-limiting toxicity of capecitabine for which no effective preventative treatment has been definitively demonstrated. This trial is conducted on the basis of preliminary data that a 3% allopurinol-based topical agent may prevent HFS.

A randomized, double-blind phase III trial will evaluate 40 patients receiving their first ever cycle of capecitabine at a dose of either 2,000 or 2,500 mg/m2 per day for 14 days. Patients will be randomly assigned to a 3% allopurinol versus a placebo cream, which will be applied to the hands and feet twice per day for 6 months after the start of capecitabine. Patients will be examined every month and the investigators will take some photographs of hands and feet. HFS toxicity grade (Common Terminology Criteria for Adverse Events [CTCAE]v3.0) will be also collected at baseline and at the end of each cycle. The primary end point is the incidence of moderate/severe HFS symptoms at the end of capecitabine treatment , based on the patient-reported dermatological exploration.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18years-old,that initiate treatment with oral capecitabine, without signs of hand-feet syndrome toxicity.
* Free acceptance to participate part in this clinical trial, with signature of the form of informed assent approved for the study, writing of the volunteer.

Exclusion Criteria:

* Age lower than 18 years
* Precedents of allergy, idiosyncrasy or hypersensitivity to the medicament.
* Denial of the patient to sign the informed assent.
* Any disorder or current / previous treatment that, in the opinion of the investigator, incapacitates the patient to take part in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-07; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Changes in the signs of hand-foot syndrome | At 1-2-3-4-5-6 months
  Erythema, descamation, vesiculation

SECONDARY OUTCOMES:
Changes in the symptoms of hand-foot syndrome | At 1-2-3-4-5-6 months
  Burning, prurigo

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona, Spain